CLINICAL TRIAL: NCT00875615
Title: Phase II Trial of Intrahepatic Artery Chemotherapy With Nexavar in Hepatocellular Carcinoma Patients
Brief Title: Cisplatin or Carboplatin and Sorafenib in Treating Patients With Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080793; SCCC-2007101; BAYER-SCCC-2007101
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Carboplatin; Cisplatin; Sorafenib

ARMS (1):
- Cisplatin or Carboplatin + Sorafenib (Experimental)
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Sorafenib

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC =6 at the investigator's discretion. Treatment is given every 6 weeks for up to 12 Cycles.
Drug: Cisplatin — Cisplatin 60 m/m² via percutaneous intrahepatic (IA) artery infusion at the investigator's discretion. Treatment is given every 6 weeks for up to 12 Cycles.
Drug: Sorafenib — Sorafenib 400 mg po bid daily starting on Day 1 (± up to 3 days) continuously.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Infusing chemotherapy directly into the liver and giving it together with sorafenib may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of infusing cisplatin or carboplatin directly into the liver and giving it together with sorafenib in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the safety of intrahepatic arterial infusion of cisplatin or carboplatin in combination with sorafenib tosylate in patients with unresectable hepatocellular carcinoma.

Secondary

* To assess the time to tumor progression in patients treated with this regimen.
* To assess the overall and progression-free survival of patients treated with this regimen.

OUTLINE: Patients receive intrahepatic arterial infusion of cisplatin or carboplatin over 30-45 minutes on day 1 and oral sorafenib tosylate twice daily on days 8-35. Treatment repeats every 42 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatocellular carcinoma (HCC) OR serum alpha fetoprotein ≥ 400 ng/mL with radiological evidence suggestive of HCC

  * Unresectable disease
* Child-Pugh class A or selected Child-Pugh class B disease (Child-Pugh score ≤ 7 points)

  * No Child-Pugh class C disease
* No disease outside the liver or macroscopic invasion of the major vessels such as the portal vein
* No known brain metastasis

  * Patients with neurological symptoms must undergo CT scan or MRI of the brain

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,000/mm³ (for patients scheduled to receive carboplatin) or ≥ 2,000/mm³ (for patients scheduled to receive cisplatin)
* Platelet count ≥ 100,000/mm³ (for patients scheduled to receive carboplatin) or ≥ 60,000/mm³ (for patients scheduled to receive cisplatin)
* Serum creatinine ≤ 1.9 mg/dL (for patients scheduled to receive carboplatin) or ≤ 1.5 mg/dL (for patients scheduled to receive cisplatin)
* Serum total bilirubin ≤ 3 mg/dL
* AST and ALT < 5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No cardiac disease, including any of the following:

  * NYHA class III-IV congestive heart failure
  * Unstable angina (anginal symptoms at rest)
  * New onset of angina within the past 3 months
  * Myocardial infarction within the past 6 months
  * Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension, defined as systolic BP > 150 mm Hg or diastolic BP > 90 mm Hg, despite optimal medical management
* No thrombolic or embolic events (e.g., cerebrovascular accident, including transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage/bleeding event ≥ CTCAE grade 2 within the past 4 weeks
* No other hemorrhage/bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* No evidence or history of bleeding diathesis or coagulopathy
* No evidence of encephalopathy
* No condition that would impair the ability to swallow whole pills
* No history of malabsorption problems
* No significant traumatic injury within the past 4 weeks
* No serious non-healing wound, ulcer, or bone fracture
* No active clinically serious infection
* No known HIV infection
* No known or suspected allergy to sorafenib tosylate or any other study agent

PRIOR CONCURRENT THERAPY:

* No prior cisplatin, carboplatin, or sorafenib tosylate
* No prior systemic chemotherapy for HCC
* No other prior systemic or locoregional therapy
* More than 4 weeks since prior major surgery or open biopsy
* No concurrent St. John's wort or rifampin

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn G. Feun, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin or Carboplatin + Sorafenib: Cisplatin : Cisplatin 60 m/m² via percutaneous intrahepatic (IA) artery infusion at the investigator's discretion. Treatment is given every 6 weeks for up to 12 Cycles.
  Sorafenib : Sorafenib 400 mg po bid daily starting on Day 1 (± up to 3 days) continuously.
  Carboplatin : Carboplatin AUC =6 at the investigator's discretion. Treatment is given every 6 weeks for up to 12 Cycles.
Period: Overall Study
Arm/Group | Cisplatin or Carboplatin + Sorafenib
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin or Carboplatin + Sorafenib
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 65 [48 to 84]
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11
Child-Pugh Score [Number; unit: participants] — Child-Pugh score is used to assess the prognosis of chronic liver disease, mainly cirrhosis. Although it was originally used to predict mortality during surgery, it is now used to determine the prognosis, as well as the required strength of treatment and the necessity of liver transplantation.
  Chronic liver disease is classified into Child-Pugh class A to C:
  Child-Pugh A: Points (5-6); 1 year survival (100%); 2 year survival (85%) Child-Pugh B: Points (7-9); 1 year survival (81%); 2 year survival (57%) Child-Pugh C: Points (10-15); 1 year survival (45%); 2 year survival (35%)
  participants
    Child-Pugh A | 10
    Child-Pugh B | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Adverse Events
Description: The number of subjects experiencing adverse events after receiving protocol therapy.
Time Frame: 36 months
Population: Of the 11 participants enrolled, 10 had results that were evaluable.
Measure: Number; unit: participants
Arm/Group | Cisplatin or Carboplatin + Sorafenib
Number analyzed (Participants) | 10
participants | 2

2. Secondary Outcome: Number of Patients Achieving Clinical Benefit
Description: Number of patients achieving complete or partial response according to RECIST criteria
Time Frame: 36 months
Population: Of the 11 participants enrolled, 10 had results that were evaluable.
Measure: Number; unit: participants
Arm/Group | Cisplatin or Carboplatin + Sorafenib
Number analyzed (Participants) | 10
participants | 6

ADVERSE EVENTS:
Arm/Group | Cisplatin or Carboplatin + Sorafenib
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin or Carboplatin + Sorafenib (N=10)
Grade 1 Diarrhea (Gastrointestinal disorders) | 2 (2)
Esophagheal Bleeding (Gastrointestinal disorders) | 1 (1) — Patient had prior history of esophageal varices.
Hemorrhoidal Bleeding (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No